CLINICAL TRIAL: NCT03546192
Title: Immunogenicity and Safety of Fluzone® Quadrivalent, Southern Hemisphere 2015 Formulation (Intramuscular Route)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC85; U1111-1143-9256 (Other: WHO)
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Results first posted 2018-08-01 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; Influenza virus vaccine; Fluzone® Quadrivalent Influenza Vaccine (No Preservative)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Participants were enrolled in two age groups: participants aged 18 to 60 years and participants aged 61 years or older.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years (Experimental): Participants aged 18 to 60 years received one 0.5-mL dose of Fluzone Quadrivalent influenza vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone Quadrivalent Influenza Vaccine
- Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older (Experimental): Participants aged 61 years or older received one 0.5-mL dose of Fluzone Quadrivalent influenza vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Fluzone Quadrivalent Influenza Vaccine — 0.5-mL, Intramuscular, SH 2015 formulation
  Other Names: Fluzone® Quadrivalent Influenza Vaccine

SUMMARY:
The aim of the study was to assess the immunogenicity and safety of Fluzone Quadrivalent influenza vaccine Southern Hemisphere (SH) 2015 formulation in participants aged 18 to 60 years as well as in participants 61 years or older.

The objectives were:

* To evaluate the compliance, in terms of immunogenicity, of the Fluzone Quadrivalent influenza vaccine SH 2015 formulation with the requirements of the European Medicines Agency (EMA) Note for guidance (NfG) CPMP/BWP/214/96
* To describe the immunogenicity of the Fluzone Quadrivalent influenza vaccine SH 2015 formulation
* To describe the safety of the Fluzone Quadrivalent influenza vaccine SH 2015 formulation

DETAILED DESCRIPTION:
All participants received 1 intramuscular dose of Fluzone Quadrivalent vaccine at the first visit.

Immunogenicity and safety were assessed in all participants. Adverse events (AE) defined in EMA NfG CPMP/BWP/214/96 were collected for 3 days after vaccination, solicited AE pre-listed in the diary card were collected for 7 days after vaccination, unsolicited AEs were collected for 21 days after vaccination, and serious adverse event (SAE) information was collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants were >= 18 years of age on the day of inclusion .
* Informed consent form had been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study.
* Self-reported thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Vaccination against influenza in the previous 12 months if administered in the context of a clinical trial or a flu vaccination campaign.
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a history of a life-threatening reaction to the vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information) .
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 3 weeks after vaccination).
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré syndrome.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion .
* Known seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, as reported by the participant. (No screening procedures were implemented.)
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38°C) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of an Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of an Investigator or employee with direct involvement in the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06-17; Primary Completion 2015-07-17 (Actual); Study Completion 2015-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Philippines (3):
  - Sanofi Pasteur Investigational Site 002, Manila
  - Sanofi Pasteur Investigational Site 003, Manila
  - Sanofi Pasteur Investigational Site 001, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Montalban C, Montellano MB, Santos J, Lavis N. Immunogenicity and safety of the 2015 Southern Hemisphere formulation of a split-virion inactivated quadrivalent vaccine. Hum Vaccin Immunother. 2018 Mar 4;14(3):593-595. doi: 10.1080/21645515.2017.1377378. Epub 2017 Oct 30. PMID 28933626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 3 centers in the Philippines from 17 June 2015 to 26 June 2015.
Pre-assignment Details: A total of 120 participants (60 for each group) were enrolled and vaccinated in the study.
Period: Overall Study
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed using the safety analysis set which included those participants who received at least 1 dose of study vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (13.9) | 68.0 (5.4) | 51.7 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 45 | 80
  Male | 25 | 15 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  Philippines | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens at Day 0 (Pre-vaccination) and Day 21 (Post-vaccination)
Description: Anti-influenza antibodies were measured using hemagglutination-inhibition (HAI) assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage. Seroprotection was defined as an antibody titer >=40 (1/dilution [dil]) at pre-vaccination and post-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: Immunogenicity analysis set included all participants who received one dose of study medication, had pre-and post-vaccination titers available and had not received vaccination against influenza in the previous 12 months if administered in the context of a clinical trial or a flu vaccination campaign.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
Participants
  A/H1N1 (Pre-Vaccination) | 41 | 37
  A/H1N1 (Day 21 Post-Vaccination) | 60 | 60
  A/H3N2 (Pre-Vaccination) | 26 | 27
  A/H3N2 (Day 21 Post-Vaccination) | 60 | 59
  B Victoria (Pre-Vaccination) | 48 | 37
  B Victoria (Day 21 Post-Vaccination) | 60 | 60
  B Yamagata (Pre-Vaccination) | 57 | 49
  B Yamagata (Day 21 Post-Vaccination) | 60 | 60

2. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies at Day 0 (Pre-vaccination) and Day 21 (Post-vaccination)
Description: Anti-influenza antibodies were measured using a HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage.
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: Analysis was performed on the Immunogenicity analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions [dil])
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
Titers (1/dilutions [dil])
  A/H1N1 (Pre-Vaccination) | 74.6 [49.9 to 112] | 48.4 [33.2 to 70.5]
  A/H1N1 (Day 21 Post-Vaccination) | 2009 [1648 to 2448] | 1083 [813 to 1442]
  A/H3N2 (Pre-Vaccination) | 27.8 [19.3 to 39.9] | 34.4 [24.6 to 48.1]
  A/H3N2 (Day 21 Post-Vaccination) | 532 [390 to 726] | 723 [525 to 994]
  B Victoria (Pre-Vaccination) | 80.0 [58.6 to 109] | 44.9 [32.3 to 62.4]
  B Victoria (Day 21 Post-Vaccination) | 1052 [849 to 1303] | 835 [654 to 1066]
  B Yamagata (Pre-Vaccination) | 209 [154 to 283] | 118 [86.0 to 161]
  B Yamagata (Day 21 Post-Vaccination) | 2242 [1828 to 2749] | 1070 [835 to 1371]

3. Primary Outcome: Geometric Mean Titer Ratio (GMTR) of Influenza Vaccine Antibodies
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage. Geometric mean titer ratio was calculated as geometric mean titer at Day 21 divided by geometric mean titer at day 0 for each specified group.
Time Frame: Day 0 (pre-vaccination), Day 21 (Post-vaccination)
Population: Analysis was performed on the Immunogenicity analysis set.
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
ratio
  A/H1N1 | 26.9 [17.1 to 42.4] | 22.4 [14.7 to 34.0]
  A/H3N2 | 19.1 [12.5 to 29.4] | 21.0 [14.0 to 31.5]
  B Victoria | 13.1 [9.72 to 17.8] | 18.6 [13.6 to 25.4]
  B Yamagata | 10.7 [7.95 to 14.5] | 9.08 [6.49 to 12.7]

4. Primary Outcome: Number of Participants With Seroconversion or Significant Increase to Influenza Vaccine Antigens
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, B Yamagata lineage. Seroconversion was defined as participants with a pre-vaccination titer <10 (1/dil) and a post-vaccination titer >= 40 (1/dil). Significant increase was defined as a pre-vaccination titer >= 10 (1/dil) and >= 4-fold increase in post vaccination titer. Number of participants with seroconversion or significant increase to Influenza vaccine antigens were reported.
Time Frame: 21 days post-vaccination
Population: Analysis was performed on the Immunogenicity analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
Participants
  A/H1N1 | 52 | 52
  A/H3N2 | 48 | 52
  B Victoria | 54 | 55
  B Yamagata | 51 | 47

5. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions
Description: A solicited reaction is an adverse event (AE) that is pre-listed in the electronic case report form (eCRF) and considered to be related to vaccination. Solicited injection site reactions: Pain (Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significantly prevent daily activity), erythema, swelling, induration, and ecchymosis (Grade 1: >=25 mm to <= 50 mm, Grade 2: >=51 to <=100 mm, Grade 3: > 100 mm). Solicited systemic reactions: Fever (Grade 1: >=38.0 degree Celsius (°C) to <=38.4°C, Grade 2: >=38.5°C to <=38.9 °C, Grade 3: >= 39°C), headache, malaise, myalgia, and shivering (Grade 1: no interference with activity, Grade 2: some interference with activity, Grade 3: significantly prevent daily activity). Number of participants with any of the Grade 1, 2 or 3 solicited injection-site and systemic reactions and Grade 3 solicited injection-site and systemic reactions were reported.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
Participants
  Any Pain | 19 | 14
  Grade 3 Pain | 0 | 0
  Any Erythema | 0 | 0
  Grade 3 Erythema | 0 | 0
  Any Swelling | 0 | 1
  Grade 3 Swelling | 0 | 0
  Any Induration | 1 | 1
  Grade 3 Induration | 0 | 0
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Fever | 1 | 1
  Grade 3 Fever | 1 | 1
  Any Headache | 8 | 3
  Grade 3 Headache | 0 | 0
  Any Malaise | 8 | 2
  Grade 3 Malaise | 0 | 0
  Any Myalgia | 6 | 4
  Grade 3 Myalgia | 0 | 0
  Any Shivering | 2 | 1
  Grade 3 Shivering | 0 | 0

6. Primary Outcome: Number of Participants Reporting Solicited Reactions Listed in the Committee for Medicinal Products for Human Use (CHMP) Note for Guidance
Description: Solicited reactions listed in the CHMP note for guidance included: injection site induration >= 50 mm for at least 4 consecutive days , injection site ecchymosis, temperature > 38.0°C for at least one day, malaise, and shivering.
Time Frame: Within 3 days after vaccination
Population: Analysis was performed on the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
Number analyzed (Participants) | 60 | 60
Participants
  Injection site induration | 0 | 0
  Injection site ecchymosis | 0 | 0
  Temperature | 0 | 1
  Malaise | 7 | 2
  Shivering | 2 | 1

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 0 (post-vaccination) up to Day 28 post vaccination .
Description: A solicited reaction is an AE that is prelisted in the eCRF and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 22/60 | 17/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone Quadrivalent Influenza Vaccine: 18 to 60 Years (N=60) | Fluzone Quadrivalent Influenza Vaccine: 61 Years or Older (N=60)
Injection Site Pain (General disorders) | 19 (19) | 14 (14)
Malaise (General disorders) | 8 (8) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.